CLINICAL TRIAL: NCT04921722
Title: Percutaneous Administration of Sirolimus in the Treatment of Superficial Complicated Vascular Anomalies: a Randomized Controlled Trial
Brief Title: Percutaneous Administration of Sirolimus in the Treatment of Superficial Complicated Vascular Anomalies
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LK210106
Record Dates: First submitted 2021-06-06; First posted 2021-06-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Kaposiform Hemangioendothelioma; Tufted Angioma; Superficial Vascular Anomalies; Superficial Lymphatic Malformations
MeSH Terms: conditions — Kaposiform Hemangioendothelioma; Tufted angioma | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical use of sirolimus (Experimental): Drop 5 ml of sirolimus oral solution and 5 g of dressing into the mixed bottle. Apply mixed gel of topical sirolimus to affected area. Use it twice a day for 6 months.
  Interventions: Drug: Percutaneous sirolimus
- Oral use of sirolimus (Active Comparator): Oral dose of sirolimus is calculated according to body surface area. Take it twice a day for 6 months. Maintain the blood concentration of sirolimus at 5-15ng/ml.
  Interventions: Drug: Oral sirolimus

INTERVENTIONS:
Drug: Percutaneous sirolimus — We compare topical and oral use of sirolimus in the treatment of superficial complicted vascular anomalies. In experimental group, we administrate percutaneous sirolimus. Drop 5 ml of sirolimus oral solution and 5 g of dressing into the mixed bottle. Apply mixed gel of topical sirolimus to affected area. Use it twice a day for 6 months.
  Other Names: Rapamycin
  Arms: Topical use of sirolimus
Drug: Oral sirolimus — We compare topical and oral use of sirolimus in the treatment of superficial complicted vascular anomalies. In active comparator group, we administrate oral sirolimus. Oral dose of sirolimus is calculated according to body surface area. Take it twice a day for 6 months. Maintain the blood concentration of sirolimus at 5-15ng/ml.
  Other Names: Rapamycin
  Arms: Oral use of sirolimus

SUMMARY:
In this study, we investigate the safety and efficacy of topical sirolimus in the treatment of superficial complicated vascular anomolies.

DETAILED DESCRIPTION:
Vascular anomaly is a kind of rare disease. According to histology, biological behavior and clinical manifestations, it can be divided into two categories: vascular tumor and vascular malformation.

mTOR inhibitors are proved with the properties of anti-proliferation and anti-angiogenesis. Therefore, they have been used in the treatment of vascular anomalies. Sirolimus, by its ability to prevent downstream protein synthesis and subsequent cell proliferation and angiogenesis, has become a novel and effective treatment. However, after the children reach complete response, there may still be skin manifestations that affect the appearance and cause psychological shadows. Therefore, intervention is required.

Studies have reported that topical sirolimus is effective in treating Kaposiform Hemangioendothelioma (KHE). It is absorbed through the skin, avoiding the first pass elimination effect of the liver. Fewer adverse reactions have been observed. In this study, we investigate the efficacy and safety of percutaneous administration of sirolimus in the treatment of superficial complicated vascular anomalies.

ELIGIBILITY:
Inclusion Criteria:

* Participant clinically or pathologically diagnosed with KHE, TA or complicated superficial vascular anomolies involving lymphatic components.

  1. The case is initial, with a relatively limited superficial lesion.
  2. The participant has residual surface lesions after oral medication.
* Participant with no use of other medication or surgical treatment
* Participant with detailed medical records of the disease at the time of screening
* Participant with signed and dated informed consent from the guardian(s)

Exclusion Criteria:

* Participants with Kasabach-Merritt Phenomenon, with platelets <50×10 9 /L.
* Participants with general disease such as hypertension, diabetes, adrenal insufficiency, neurological diseases, liver and kidney dysfunction, and cardiopulmonary insufficiency.
* Participants with other hematological diseases or solid tumor.
* Participants allergic to sirolimus or dressing.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Effective rate | From admission to follow-up six months
  Achauer BM et al. made the four-level standard as follows. Grade I: tumor size and skin lesion color regression ≤ 25%; grade II: tumor size and skin lesion color regression 25%-50%; grade III: tumor size and skin lesion color regression 50-75%; grade IV: tumor size and skin lesion color regression ≥75%. After 6 months of treatment, the pzrticipant will be evaluated. Grade I will be viewed as invalid. Grade II and grade III will be viewed as effective, and grade IV will be viewed as very effective. Those in grade Ⅱ, Ⅲ or Ⅳ will be calculated in effectiveness rate.

SECONDARY OUTCOMES:
Changes of resistance coefficient | From admission to follow-up six months
  Measured by ultrosonic doppler flowmetery at follow-up
Incidence of adverse events | From admission to follow-up six months
  Adverse events will be reported according to Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v4.0). Incidence of complications such as oral ulcers, abnormal liver enzymes, infections will be recorded. It is defined as occurring if individual subject has any of the above complications during the 6-month intervention
Platelet count | From admission to follow-up six months
  Platelet count is one of the major indicators of response to treatment. It is supposed to be greater than 100×10^9/L.
Changes of peak blood flow | From admission to follow-up six months
  Measured by ultrosonic doppler flowmetery at follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China